CLINICAL TRIAL: NCT03577886
Title: A Phase 1 Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of CDX-6114 Following Single, Ascending Oral Dose Administration to Healthy Volunteers.
Brief Title: Safety and Tolerability of CDX-6114 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Codexis Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDX6114-001
Record Dates: First submitted 2018-06-14; First posted 2018-07-05 (Actual); Last update posted 2018-09-20 (Actual); Status verified 2018-07

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Dose-escalating, Randomized, Double-blinded, Placebo-controlled.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CDX-6114 (Experimental): 0.225, 0.75, 2.25 and 7.5 g
  Interventions: Drug: CDX-6114
- Placebo (Placebo Comparator): Phosphate Buffer Diluent solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CDX-6114 — CDX-6114 will be administered as a single, oral dose solution at dose levels of 0.225, 0.75, 2.25, and 7.5 g.
  Arms: CDX-6114
Drug: Placebo — Phosphate Buffer Diluent oral solution
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and tolerability of an oral solution of CDX-6114 when administered as a single dose in healthy volunteers.

DETAILED DESCRIPTION:
This is a Phase 1, double-blind, placebo-controlled study in approximately 32 healthy volunteers who are 18 to 55 years old. Four cohorts are planned, each consisting of 8 subjects; the cohorts as planned are 0.225, 0.75, 2.25, and 7.5 g in oral solution. Increasing doses of CDX-6114 will be assessed sequentially until the final dose is evaluated or any of the stopping criteria are reached. Subjects will each receive a single dose and then will be followed for a total of 22 days (3 weeks).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female, non-smoking, subjects between the ages of 18 and 55 years, inclusive, at the time of screening.
2. Have a body mass index (BMI) between 18.0 and 30.0 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive.
3. Good general health, as determined by an experienced physician based on a medical evaluation including detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead electrocardiogram (ECG), neurological assessment and clinical laboratory tests.
4. Male subjects and their female spouse/partner(s) who are of childbearing potential:

   1. Must agree to stay abstinent (where abstinence is the preferred and usual life-style of the subject), starting at screening and continuing throughout the clinical study period, and for 90 days after study drug administration.

      Or
   2. Must be using highly effective contraception consisting of 2 forms of birth control (1 of which must be a barrier method) starting at screening and continuing throughout the clinical study period, and for 90 days after study drug administration.
   3. These requirements do not apply to participants in a same sex relationship.
5. Male subjects must agree not to donate sperm starting at screening and continuing throughout the clinical study period, and for 90 days after study drug administration.
6. Female subjects of childbearing potential:

   1. Must agree not to become pregnant during the clinical study period and for 30 days after study drug administration.
   2. Must have a negative serum pregnancy test at screening.
   3. If heterosexually active, must agree to consistently use a form of highly effective birth control, in combination with a barrier method starting at screening and continuing throughout the clinical study period, and for 30 days after study drug administration

      Or
   4. Must agree to stay abstinent (where abstinence is the preferred and usual life-style of the subject), starting at screening and continuing throughout the clinical study period, and for 30 days after study drug administration.
   5. These requirements do not apply to participants in a same sex relationship.
7. Female subjects of non-childbearing potential:

   1. Must have a confirmed clinical history of sterility

      Or
   2. Must be postmenopausal as defined as: amenorrhea for at least 1 year prior to screening and a laboratory confirmed serum follicle stimulating hormone (FSH) level ≥ 40mIU/mL.
8. Female subjects must agree not to breastfeed starting at screening and continuing throughout the clinical study period, and for 90 days after study drug administration.
9. Female subjects must agree not to donate ova starting at screening and continuing throughout the clinical study period, and for 90 days after study drug administration.
10. Subject must be competent to understand the nature of the study & capable of giving written informed consent. Be willing to report for the scheduled study visits and communicate to study personnel about adverse events and concomitant medication use.
11. Subject must abstain from the following foods from 1 week prior to study drug administration until the last PK sample has been obtained: grapefruit juice or products, pomegranate juice or products, foods containing poppy seeds, and/or drinks or foods containing quinine (e.g., tonic water) or Seville oranges (e.g. orange marmalade).
12. Subject agrees not to participate in another interventional study while participating in the present clinical study.

Exclusion Criteria:

1. Female subject who has been pregnant within the 6 months prior to screening or breastfeeding within the 3 months prior to screening.
2. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies and childhood asthma) at time of screening or study drug administration.
3. Current or chronic history of gastrointestinal disorders or conditions interfering with normal gastrointestinal anatomy or motility. Examples include gastrointestinal bypass surgery, cholecystectomy, partial or total gastrectomy, gastric band surgery, small bowel resection, vagotomy, malabsorption, Crohn's disease, ulcerative colitis, irritable bowel syndrome (IBS) or celiac sprue.
4. Treatment with any anti-platelet and/or anticoagulant medication.
5. Evidence or history of specific food intolerance. Examples include gluten intolerance, lactose intolerance, or dairy food intolerance or any food/ingredient included in the standard protein breakfast.
6. A positive result, on screening, for serum hepatitis B surface antigen (HBsAg), hepatitis A virus antibodies (HAV), hepatitis C virus antibodies (HCV) or antibodies to human immunodeficiency virus type 1 (HIV-1) and/or type 2 (HIV-2).
7. A positive pre-study drug/alcohol screen. However, there is the option to re-screen during the screening period at the discretion of the Principal Investigator (PI) or delegate in the case of a positive pre-study drug screen for a prescribed medication e.g. codeine.
8. Subject has a history of drinking > 21 units of alcohol/week for male subjects or > 14 units of alcohol/week for female subjects within the 3 months prior to screening.
9. Subject has a history of regular smoking (daily or most days in a week) or the use of nicotine products (3 or more nicotine-containing products) within the 6 months prior to screening.
10. Subject has used any recreational drugs of abuse within the 3 months prior to screening.
11. Subject has a pulse rate <40 or > 100 bpm; mean systolic blood pressure (SBP) > 140 mmHg; mean diastolic blood pressure (DBP) > 90 mmHg at screening. Repeat measurements are allowed at the discretion of the PI or delegate.
12. Subject has any clinically significant abnormalities at screening in rhythm, conduction or morphology of the resting ECG and any clinically significant abnormalities in the 12-lead ECG, as considered by the Investigator, that may interfere with the interpretation of QTc interval changes including abnormal ST-T wave morphology.
13. Subject has prolonged QTcF (QT interval corrected for heart rate using Fridericia's formula) > 450 ms for male subjects or > 470 ms for female subjects, or a shortened QTcF < 300 ms or a family history of prolonged QT syndrome, at screening.
14. Subject has any clinically significant abnormalities in clinical chemistry, hematology, or urinalysis at screening as judged by the Investigator, including: Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), alkaline phosphatase (ALP), gamma glutamyl transferase (GGT) or Total bilirubin (TBL) up to 1.5 times above the Upper Limit of Normal (ULN).
15. Plasma donation within the 14 days prior to screening or any whole blood donation/significant blood loss > 500 mL during the 3 months prior to screening.
16. Treatment with any Investigational Drug or Device/Treatment within the 30 days prior to the administration of study drug.
17. Use of any prescribed or non-prescribed medication including herbal and dietary supplements, antacids, analgesics (other than oral contraceptives, paracetamol or multi-vitamins) during the two weeks prior to the administration of the study drug, or up to a minimum of 5 times the half-life of the medication if it has a long half-life.
18. Exposure to more than four new chemical entities within the 12-month period prior to the administration of the study medication.
19. Known allergy or adverse reaction history to any of the oral dose formulation components e.g. mannitol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2018-07-04 (Actual); Primary Completion 2018-08-21 (Actual); Study Completion 2018-09-04 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure of the study will be the incidence of treatment-emergent Adverse events experienced by the Subjects following oral administration of CDX-6114 | Up to 22 days after drug administration
  Will be measured by assessing the frequency and the nature of the AE's reported

SECONDARY OUTCOMES:
Pharmacokinetics of CDX-6114, | Up to 24 hours after drug administration
  Assessed by the serum levels of CDX-6114 following oral administration of CDX-6114
Pharmacodynamics of CDX-6114 | Up to 24 hours after drug administration
  Assessed by the plasma levels of Phenylalanine and Cinnamic acid following oral administration of CDX-6114.

CONTACTS AND LOCATIONS:
Overall Officials: Sam Salman, Principal Investigator — Linear Clinical Services
Locations (1):
- Linear Clinical Services, Perth, Western Australia, Australia

IPD SHARING:
Plan to Share IPD: No